CLINICAL TRIAL: NCT03839251
Title: Effectiveness of Aripiprazole Long-acting Injection in Recent Onset and Chronic Schizophrenia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Young Chul Chung, Professor of Psychiatry, Chonbuk National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUH 2018-02-011-005
Record Dates: First submitted 2019-01-29; First posted 2019-02-15 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Schizophrenia
Keywords: aripiprazole; long-acting injection
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- abilify maintena (Other): aripiprazole 400mg or 300mg, IM, Once a month
  Interventions: Drug: abilify maintena

INTERVENTIONS:
Drug: abilify maintena — aripiprazole 400mg or 300mg, IM, Once a month
  Other Names: aripiprazole

SUMMARY:
The aim of the study is to investigate the effectiveness of Aripiprazole long-acting injection in recent onset and chronic schizophrenia patients

DETAILED DESCRIPTION:
The aim of this study is to investigate the effectiveness of Aripiprazole long-acting injection in recent onset and chronic schizophrenia patients

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia according to DSM-5 diagnostic standards
* men and women aged 19 and under 60
* a person who is being given an atypical antipsychotic.
* Patients should be able to reasonably cooperate with the questionnaire to be used for the study
* a person who fully understands the purpose of the study and signs the consent
* stable outpatient before screening without changing the volume of antipsychotics for at least two weeks

Exclusion Criteria:

* a person who has a serious and unstable physical condition either now or in the past
* A fertile woman who is currently pregnant or breastfeeding, or who is either unwilling or unable to use acceptable contraception until the clinical trial is complete.
* a person suffering from severe drug allergies or complex and severe drug reactions
* Patients who have taken clozapine in the last 60 days
* subjects showing significant risk of suicide or significant risk of violent behavior based on past history or investigator's judgment

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline PSP(Personal and Social Performance scale) at 12weeks | 12weeks
  PSP(Personal and Social Performance scale) was measured in baseline and 12week. Minimum of PSP(Personal and Social Performance Scale) is 1, maximum is 100. The lower number is worse outcome.
Change from Baseline PSP(Personal and Social Performance scale) at 24weeks | 24weeks
  PSP(Personal and Social Performance scale) was measured in baseline and 24week. Minimum of PSP(Personal and Social Performance Scale) is 1, maximum is 100. The lower number is worse outcome.

SECONDARY OUTCOMES:
Efficacy Assessment by CGI-S(Clinical global impression-schizophrenia) | baseline, 4weeks, 8weeks, 12weeks, 16weeks, 20weeks, 24weeks
  Clinical global impression-schizophrenia(CGI-S)
  There are Positive Symptoms, Negative Symptoms, Depressive Symptoms, Cognitive Symptoms and Overall severity in the Clinical global impression-schizophrenia(CGI-S). minimum of each items(Positive Symptoms, Negative Symptoms, Depressive Symptoms, Cognitive Symptoms and Overall severity) is 1, Maximum is 7. The higher number is worse outcome.
Efficacy Assessment by ERT(Emotional Recognition Test) | baseline, 24weeks
  Emotional Recognition Test(ERT)
  minimum of ERT(Emotional Recognition Test) total score is 0, Maximum is 54. The lower number is worse outcome.
Efficacy Assessment by PANSS(Positive and Negative Syndrome Scale) | baseline, 12weeks, 24weeks
  Positive and Negative Syndrome Scale(PANSS)
  There are Positive Scale, Negative Scale and General Psychopathology Scale in the PANSS(Positive and Negative Syndrome Scale). minimum of each items(Positive Scale, Negative Scale and General Psychopathology Scale) is 1, Maximum is 7. The higher number is worse outcome.
Efficacy Assessment by self rating scale | baseline, 12weeks, 24weeks
  Subjective Wellbeing under Neuroleptics(SWN-K)
  SWN-K(Subjective Wellbeing under Neuroleptics) consists of 20 questions. The minimum score for each question is zero and the maximum score is five. The reverse scoring questions include 1,4,6,9,10,11,12,14,16,17. The total score of the whole item is obtained, and the lower the score, the worse the subjective well-being.
Safety Assessment by Simpson-Angus Scale(SAS) | baseline, 12weeks, 24weeks
  Simpson-Angus Scale(SAS)
  minimum of each items(Gait, Arm Dropping, Shoulder Shaking, Elbow Rigidity, Fixation of Position or Wrist Rigidity, Leg Pendulousness, Head Dropping, Glabella Tap, Tremor, Salivation) in the SAS(Simpson-Angus Scale) is 0, Maximum is 4. minimum of total scores in the SAS(Simpson-Angus Scale) is 0, Maximum is 40. The higher number is worse outcome.
Safety Assessment by Barnes Akathisia Rating Scale(BARS) | baseline, 12weeks, 24weeks
  Barnes Akathisia Rating Scale(BARS)
  minimum of each items(Objective, Subjective, Distress related to restlessness) in the BAS(Barnes Akathisia Rating Scale) is 0, Maximum is 3. Minimum of Global clinical assessment of akathisia in the BARS is 0, Maximum is 5. The higher number is worse outcome.
Safety Assessment by Abnormal Involuntary Movement Scale(AIMS) | baseline, 12weeks, 24weeks
  Abnormal Involuntary Movement Scale(AIMS)
  minimum of each items in the AIMS(Abnormal Involuntary Movement Scale) is 0, Maximum is 4. The higher number is worse outcome.
Safety Assessment by self report scale | baseline, 12weeks, 24weeks
  Visual Analogue Scale(VAS)
  minimum of VAS(Visual Analogue Scale) is 0, Maximum is 10. The higher number is worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Young-chul Chung, MD, Principal Investigator — Chonbuk National University Hospital
Locations (5):
- South Korea (5):
  - Department of Psychiatry, Inje University Haeundae Paik Hospital, Busan
  - Department of Psychiatry, Kyungpook National University Hospital, Daegu
  - Department of Psychiatry, Yeungnam University Medical Center, Daegu
  - Department of Psychiatry, Chonnam National University Medical School, Gwangju
  - Department of Psychiatry, Chonbuk National University Hospital, Jeonju